CLINICAL TRIAL: NCT04078347
Title: Changes of Skin Temperature for Evaluation of Paravertebral Block: A Prospective Observational Study Using Infrared Thermography
Brief Title: Infrared Thermography to Evaluate the Effect of Paravertebral Block
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, Vice Director, Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: TJ-IRB20190424
Record Dates: First submitted 2019-08-06; First posted 2019-09-06 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-11

CONDITIONS: Paravertebral Block
Keywords: Paravertebral block; Infrared thermography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Successful Paravertebral block: Pinprick test was evaluated at 20 min after Paravertebral block. Pinprick sensation was assessed using a 22-gauge short bevel needle from T2 to T10 at midclavicular line bilaterally . Pinprick response was recorded quantitatively as 1 (sensation) or 0 (no sensation/numb). Successful block was defined as the pinprick score was 0 at 20 min after block. Otherwise, it was defined as a failed block.
  Interventions: Procedure: Paravertebral block at T4 and T5 level
- Failed Paravertebral block: Pinprick test was evaluated at 20 min after Paravertebral block. Pinprick sensation was assessed using a 22-gauge short bevel needle from T2 to T10 at midclavicular line bilaterally . Pinprick response was recorded quantitatively as 1 (sensation) or 0 (no sensation/numb). Successful block was defined as the pinprick score was 0 at 20 min after block. Otherwise, it was defined as a failed block.
  Interventions: Procedure: Paravertebral block at T4 and T5 level

INTERVENTIONS:
Procedure: Paravertebral block at T4 and T5 level — Paravertebral block is performed at T4 and T5 level under realtime ultrasound guidenance with 10ml of 0.5% ropivacaine for each block, respectively.

SUMMARY:
The aim of this prospective observational study was to evaluate the changes of skin temperature after the paravertebral block measured by infrared thermography.

DETAILED DESCRIPTION:
Methods: Patients scheduled for elective surgery with paravertebral block will receive infrared thermography measures 5 min before the block and continous to 20 min after the block. The sensitivity, specificity of infrared thermography as diagnostic methods will be determined by receiver operator characteristic analysis.

ELIGIBILITY:
Inclusion Criteria:

* With informed consent
* American Society of Anesthesiologists physical status Ⅰ-Ⅱ
* Undergo elective surgery with planned paravertebral block

Exclusion Criteria:

* Refusal to participate in the study
* pre-existing infection at the block site
* younger than 18-yr-old
* BMI>35
* significant thoracic kyphoscoliosis
* Those who had taken vasodilatory drugs before surgery
* history of previous thoracic or breast surgery
* Preoperative analgesic medications
* Any contraindications to peripheral nerve block such as coagulation abnormalities, allergy to local anaesthetics, peripheral neuropathy.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery with planned paravertebral block for multimodel analgesia.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Changes of skin temperature | From baseline up to 20 minutes after block
  Changes of skin temperature determined by infrared thermography

SECONDARY OUTCOMES:
Noinvasive blood pressure | From baseline up to 20 minutes after block
  Vital signs
Heart rate | From baseline up to 20 minutes after block
  Vital signs
SPO2 | From baseline up to 20 minutes after block
  vital signs
Sensory block level | From baseline up to 20 minutes after block
  Sensory block level determined by pinprick.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Mei, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
For patient's privacy

REFERENCES:
- [Derived] Zhang S, Liu Y, Liu X, Liu T, Li P, Mei W. Infrared thermography for assessment of thoracic paravertebral block: a prospective observational study. BMC Anesthesiol. 2021 Jun 11;21(1):168. doi: 10.1186/s12871-021-01389-4. PMID 34116642